CLINICAL TRIAL: NCT00748774
Title: Primary Brain Tumor Patient and Caregiver Congruence in Symptom Report Using the M.D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT)
Brief Title: Brain Tumor Patient-Caregiver Congruence, MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0117
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Brain Tumor
Keywords: Primary Brain Tumor; Caregivers; Symptom Severity; Questionnaire; M.D. Anderson Symptom Inventory-Brain Tumor; MDASI-BT
MeSH Terms: conditions — Brain Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDASI-BT: MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) questionnaire given to patients with a primary brain tumor and their caregivers.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Two questionnaires taking about 10 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this study is to compare patient ratings of how severe their own symptoms may be, with their caregivers' ratings of how severe they think the patients' symptoms may be. This will be compared using a questionnaire that is given to patients with brain tumors and their caregivers.

Researchers will also study any effects that these patients' neurocognitive function may have on these patients' and their caregivers' ratings of how severe the brain cancer symptoms may be.

DETAILED DESCRIPTION:
Study Visit:

If you and your caregiver agree to take part in this study, you will both complete 2 questionnaires. You will be in separate rooms when you complete the questionnaires.

The first questionnaire is a demographic questionnaire that asks basic questions such as your age and employment status.

Your second questionnaire asks about any brain cancer symptoms that you may be experiencing, and asks you to rate how severe they may be.

Your caregiver's second questionnaire asks the same questions as yours. It asks the caregiver to rate how severe he or she believes your symptoms may be.

In total, the questionnaires should take about 10 minutes to complete.

Symptom Review:

The study staff will review the questionnaire responses right away. If you rate any symptom as severe as 7 or higher, the study staff will tell you to contact your doctor who is treating the cancer. The study staff will also contact your doctor who is treating the cancer. Otherwise, your questionnaire responses will only be used for research and there are no plans to contact your doctor.

Length of Study Participation:

After you and your caregiver complete the questionnaires this one time, your and your caregivers' active participation in this study will be over.

The study chair will also collect information from your medical record. This information will include your medical history and the results of the neurocognitive testing (routine tests of "thinking" skills such as your memory and concentration).

This is an investigational study. Up to 120 patients and 120 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging consistent with a primary brain tumor or prior pathologic diagnosis of primary brain tumor
2. Referred for neurocognitive function testing as part of the plan of care
3. Age > or = 18 years of age
4. Ability to speak, read, and write the English language
5. Caregiver Attribute: Identified by the patient as being primarily involved in the patients' care in the home setting (biologic, legal, or functional relationship)
6. Caregiver Attribute: Able to speak, read, and write the English language
7. Both patient and caregiver have to agree to participate
8. The caregiver needs to be present at the time the patient is recruited

Exclusion Criteria:

1. Patients less than 18 years of age will be excluded from this study.
2. Patients will be excluded from the study if they are unable to complete the self-report questionnaire or participate in neurocognitive testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with a brain tumor who are going to have neurocognitive testing as part of routine care and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mean Caregiver Ratings of Symptom Severity (using the mean of all the items from the MDASI-BT) in Patient-Caregiver Dyads | Participant involvment is 10 minutes to complete MDASI-BT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org